CLINICAL TRIAL: NCT02293590
Title: An Open Label, Randomised Study to Compare the Efficacy of Certolizumab Pegol (CZP) Plus a Dynamic or Fixed Dose Treatment Strategy in Patients With Rheumatoid Arthritis, a Phase II Study
Brief Title: RICE: Remission by Intra-articular Injection Plus CErtolizumab
Acronym: RICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rüdiger B. Müller (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Rüdiger B. Müller, Dr. med. Rüdiger Müller, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKSG13/104/2B
Record Dates: First submitted 2014-10-30; First posted 2014-11-18 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab pegol; DMARD; Joint injection; Glucocorticoids
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Sulfadiazine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intensive, adapted treatment strategy (Experimental): Experimental: intensive, adapted treatment strategy Certolizumab pegol (CZP, Cimzia (R)): 200mg every 2 weeks after loading d 400mg at Weeks 0, 2 and 4
  DMARD:
  Patients without sufficient treatment response will be taken to the next step according to the therapeutic algorithm or next drug, for example: 15=>25mg Metoject (R)/week => Leflunomide Gebro (R)20mg/d => Salazopyrine EN(R) 2000mg/d
  Glucocorticoids:
  At Week, 0 patients will be initiated on Spiricort (R) 20mg/d and tapered every 5 days
  Joint injections:
  Starting at Week 0 up to 5 joint injections may be conducted into synovitic joints at every visit of the study.
  The maximum cumulative Lederlon (R) dose is 100mg/visit. Joints are to be infiltrated with the following doses of triamcinolone and lidocaine
  Interventions: Drug: Certolizumab Pegol
- fixed-dosed program (Active Comparator): Intervention:
  Certolizumab pegol (Cimzia (R), CZP) CZP of 400mg at Weeks 0, 2 and 4, followed by 200mg injections from Week 6, every 2 weeks until Week 24.
  DMARD:
  Patients are to continue to receive their stable weekly dose of DMARD as noted at study entry for the duration of the study (24 weeks)
  Glucocorticoids:
  Prednisolone (Spiricort (R)) daily dose of ≤ 10 mg
  Joint injections:
  None
  Interventions: Drug: Certolizumab Pegol

INTERVENTIONS:
Drug: Certolizumab Pegol
  Other Names: Cimcia; Methoject; Lederlon; Leflunomid Gebro; Salazopyrin EN; Spiricort; Xyloneural

SUMMARY:
Tight control of an adaptive concomitant treatment strategy after initiation of CZP will lead to an improved outcome of RA patients with an active disease despite DMARD treatment.

DETAILED DESCRIPTION:
Certolizumab pegol (CZP) is a tumor necrosis factor (TNF) antagonist which is marketed for the treatment of moderate to severe rheumatoid arthritis (RA) (Keystone, 2008) when given in combination with methotrexate (MTX). CZP is a PEGylated Fab' fragment of humanized anti-TNF antibody with a high affinity for TNF.

RA is a chronic inflammatory autoimmune disease with multiple treatment strategies and combination therapies available including analgesia, anti-inflammatory drugs and disease-modifying anti-rheumatic drugs. Previous trials have demonstrated positive results from the use of CZP but have compared its use to placebo in a fixed dose concomitant medication regime rather than using a more realistic dynamic treatment strategy normally employed in the clinical outpatient care of RA.

This trial is aimed at comparing the use of CZP in patients with moderate to severe RA when administered in conjunction with an intensive, adapted treatment strategy (Group A) versus a fixed-dosed program (Group B). CZP will be given in conjunction with MTX (a disease modifying anti-arthritic drug - or DMARD), steroidal therapy in the form of prednisolone and joint infiltrations of triamcinolone (another corticosteroid) and lidocaine (a pain therapy). Both treatment arms will include these concomitant medications but there will be an intensive adaptive approach adopted for the 'treat to target' population of Group A with a more fixed-dose approach set-out for Group B. Patients will be centrally randomized after screening to ensure a 50:50 ratio for both Groups in the study.

STUDY HYPOTHESIS

Tight control of an adaptive concomitant treatment strategy after initiation of CZP will lead to an improved outcome of RA patients with an active disease despite DMARD treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older at the time of consent
2. Able to give informed consent
3. Patients diagnosed as having established and active rheumatoid arthritis classified according to the 2010 American College of Rheumatology/European League against Rheumatism (ACR/EULAR) criteria (Aletaha D et al 2010) for a period of ≥ 3 months counting from the first DMARD treatment initiated. Active rheumatoid arthritis is characterised as all of the following:

   * ≥6 tender joint out of the 68 joint count
   * ≥6 swollen joints out of the 66 joint count
   * ESR ≥ 20mm/h or CRP ≥7mg/l
4. Has a been found to be intolerant to, or had an inadequate clinical response to at least 1 DMARD
5. Is currently being treated with DMARDs for ≥ 12 weeks and has reached a stable dose for ≥ 4 weeks.
6. Is currently receiving a corticosteroid (e.g. prednisolone or equivalent) and has reached a stable dose of ≤ 10mg/d for ≥ 4 weeks (patients without current corticosteroid treatment for ≥ 4 weeks may also be included.
7. Available for the whole duration of the study.
8. Female subjects of childbearing potential must use maximally effective birth control during the period of therapy, must be willing to use contraception for the duration of the study (starting from randomisation and ending up to Week 24 at Day 168/Safety follow-up visit). Must have a negative pregnancy test upon entry into the study. Otherwise, female subjects must be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile.
9. Male subjects must be surgically sterile or willing to use a double barrier contraception method upon enrolment, for the duration of the study (starting from randomisation and ending up to Week 24 at Day 168/Safety follow-up visit).

Exclusion Criteria:

1. Pregnant or breastfeeding women or such with a child-bearing potential who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the entire study period (up to Week 24 at Day 168/Safety follow-up visit)
2. Subjects with a history of cancer in the last 5 years, or with a current screening suspicious for cancer, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ
3. Subjects with evidence of untreated, active or latent bacterial (e.g. tuberculosis) or viral infections (e.g. Human Immunodeficiency Virus (HIV), Hepatitis B or C) at the time of potential enrolment
4. Subjects with any serious bacterial infection within the last 3 months, unless treated and resolved with antibiotics, or any untreated, chronic bacterial infection
5. Having participated in another drug or an interventional study within 30 days preceding the present study screening
6. Any previous treatment with CZP
7. Any previous treatment with a biological DMARD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
To assess the percentage of study participants achieving American College of Rheumatology 50% (ACR50) clinical response by the Week 24 assessments | 24 weeks
  Efficacy rates as measured by the percentage of study participants achieving American College of Rheumatology 50% (ACR50) clinical response by the Week 24

SECONDARY OUTCOMES:
To compare the efficacy rates of CZP between the two treatment groups following 8, 12, 18 and 24 weeks of treatment | 8, 12, 18 and 24 weeks
  Efficacy rates as measured by ACR20/50/70 at weeks 8, 12, 18 and 24 weeks to determine the % of treatment responders in each study Group over the study period.
To compare the proportion of patients reaching either a low disease activity status (LDAS) or a full remission of their RA across both treatment groups at weeks 8, 12, 18 and 24 | weeks 8, 12, 18 and 24
  Efficacy rates as measured by patients achieving Low DAS is defined (LDAS) or a full clinical remission according to the EULAR at weeks 8, 12, 18 and 24 weeks. LDAS as a DAS-28 score of less than 3.2. The DAS-28 is defined by the number of tender and swollen joints calculated from 28 joints mainly from the upper limbs, the ESR and the patient's global assessment of disease activity.
  Remission will be defined as a DAS-28 score of less than 2.6 and/or according to the Boolean definition of remission (Felson 2011): swollen joint count, tender joint count, patients' global assessment of disease activity, CRP (mg/dl) all ≤1*
To compare the relative time taken for patients to reach remission across the two treatment groups | weeks 8, 12, 18 and 24
  Efficacy rates as measured by the average number of weeks of treatment required for patients to reach remission of their RA. Clinical remission to be evaluated via the EULAR and DAS-remission criteria
To compare the cumulative corticosteroid dose for patients across the two study treatment groups following 24 weeks of treatment | 24 weeks
  Efficacy as calculated of the cumulative corticosteroid dose for patients completing the 24 week study period across the two treatment groupsCalculation of the cumulative corticosteroid dose for patients completing the 24 week study period across the two treatment groups
To compare the safety and tolerability of CZP between the two treatment groups following 8, 12, 18 and 24 weeks of treatment | 8, 12, 18 and 24 weeks
  Safety as calculated by the occurrence of treatment emergent adverse event (TEAE, adverse events occurring after baseline of the study) across the two treatment groups
To conduct pharmacokinetic analysis to compare the CZP serum levels following 24 weeks of treatment across both of the treatment groups | 24 weeks
  Efficacy analysis as analysed by a pharmacokinetic assessments are to be conducted at Visit 3/week 4 (day 28) and visit 7/Week 24 (Day 168 post initiation of CZP treatment)
To compare the development of anti-CZP antibodies following 24 weeks of treatment across both of the treatment groups | 24 weeks
  Efficacy analysis as analysed two single timepoint anti-CZP antibody assessments are to be conducted at Visit 2/Week 0 and Visit 7/Week 24 (Day 168 post initiation of CZP treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Rueediger B Mueller, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Kantonsspital St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland